CLINICAL TRIAL: NCT00994201
Title: Pilot Study of DCE-MRI, DW-MRI, and MRS in the Assessment of Head and Neck Cancer Response to Chemo-radiation
Brief Title: Magnetic Resonance Imaging (MRI) in the Assessment of Head and Neck Squamous Cell Carcinoma (HNSCC) Response
Status: Terminated | Type: Observational
Why Stopped: Study never accrued sufficient subjects
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Medical Research Foundation, Oregon (Other); Radiological Society of North America (Other)
Responsible Party: Principal Investigator, James Tanyi, Clinical Associate Professor, OHSU Knight Cancer Institute
Other Study IDs: OHSU IRB00005554
Record Dates: First submitted 2009-10-13; First posted 2009-10-14 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: DCE-MRI, DW-MRI and MRS — Patients will undergo Dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI), Diffusion-weighted magnetic resonance imaging (DW-MRI), Magnetic resonance spectroscopy (MRS) prior to the initiation of chemoradiation and before their second cycle of chemotherapy.
  Healthy volunteers will undergo DCE-MRI, DW-MRI and MRS.

SUMMARY:
The purpose of this study is to see if new techniques of measuring HNSCC tumors with magnetic resonance imaging (MRI) can help predict how well the tumors will respond to combined chemotherapy and radiation treatment. The investigators hope to find a reliable method to determine whether or not a patient's cancer is responding to chemo-radiation early in their treatment using an MRI, such that that cancer treatments could be tailored to the individual more effective in the future. The MRI techniques include dynamic contrast-enhanced magnetic resonance imaging (DCE-MRI), diffusion-weighted magnetic resonance imaging (DW-MRI), and magnetic resonance spectroscopy (MRS). Participants will be subjected to two sessions of MRI scans: one before the initiation of their regular treatment and the second before their second cycle of chemotherapy. Each scanning session will last approximately 45 minutes.

DETAILED DESCRIPTION:
DCE-MRI, DW-MRI, MRS have the potential to measure early cellular changes that occur in response to successful therapies, such as chemoradiation, and have been demonstrated to be early predictors not only of therapeutic response, but also of overall survival for other malignancies. Our long-term goal is to use these imaging techniques to develop non-invasive functional imaging methodologies that would be better predictors of pathological response than the current clinical standard.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of loco-regionally advanced (stage III or IV) squamous cell carcinoma of the head and neck (oropharynx, hypopharynx and larynx)
* Age > 18 years
* No prior surgery, chemotherapy or radiation therapy for head and neck cancer
* Scheduled to receive chemoradiation for definitive therapy

Exclusion Criteria:

* Contraindications to MRI (pacemaker, aneurysm clip, mechanical and/or electrical device or metallic fragment, severe claustrophobia)
* Contraindications to gadolinium
* Severe, active co-morbidity
* Major medical illnesses or psychiatric impairments
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be recruited by the Oregon Health and Science University head and neck oncology staff.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Determination of early or a prior prognostic markers of head and neck cancers, as measured by DCE-MRI, DW-MRI, and MRS, that characterize the differences between clinical responders and non-responders. | September 2011

SECONDARY OUTCOMES:
Correlation between early/a prior marker and progression-free survival. | September 2011

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tanyi, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: Oregon Health and Science University — http://www.ohsu.edu